CLINICAL TRIAL: NCT02267187
Title: Structural Fat Grafting for Craniofacial Trauma Using Manual Technique for Processing Fat Graft Material
Acronym: BTI++
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, J. Peter Rubin, MD, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO14040197
Record Dates: First submitted 2014-08-08; First posted 2014-10-17 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Facial Injuries
Keywords: Craniomaxillofacial (CMF); Battle-injured (BI); Facial Trauma; Fat Grafts; Autogenous Fat Transfers (AFT); Wounded Warriors
MeSH Terms: conditions — Facial Injuries | interventions — Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fat Graftting (Experimental): For the purpose of this study the fat grafting procedure is a research procedure. It is very important to note that this research procedure is not an experimental procedure. Fat grafting is a minimally invasive clinical procedure that has been widely used by plastic surgeons within reconstructive surgery for many years. Fat grafting is known as a filler providing an accurate means to restoring facial soft tissue structure.
  Interventions: Procedure: Fat Grafting; Drug: General Anesthesia; Device: Coleman Cannulas; Other: Tefla non-adherent gauze pad

INTERVENTIONS:
Procedure: Fat Grafting — Fat Grafting is a procedure that involves moving a person's own fat from an area of the body where it is less needed to another area of the body to improve its appearance. The fat is usually taken from the thighs or abdomen with a small liposuction tube and then moved to an area that has lost volume or fullness due to aging, trauma, surgery, birth defects, or other causes.
Drug: General Anesthesia — A medicine that will relax and assist the subject in keeping unconscious (in a sleep like state) during the entire procedure.
Device: Coleman Cannulas — The plastic surgeon, will use small narrow tube-like instruments called cannulas, will remove fat from various places throughout the body (commonly the abdomen and thighs). The plastic surgeon will then use the Coleman cannulas (specialized smaller cannulas with varied shapes and tip sizes specifically made to deliver smaller amounts of fat) to fill the desired area.
Other: Tefla non-adherent gauze pad — The processing of the fat graft material is done using a Tefla non-adherent gauze pad in a rolling technique that separates the aqueous and oil layers from the injected component.

SUMMARY:
This study will examine the impact of the fat grafting procedure on facial appearance and quality of life over time by precisely measuring soft tissue volume with CT scans, assessing appearance with 2D and 3D photography and standard photography and evaluating quality of life through various validated psychosocial measures. This study will be a very important evaluation of the effectiveness of this therapy, and will help guide clinicians in applying this technique. Additionally, laboratory testing of the injected fat material will be performed so that the results may be correlated with clinical outcomes in the future.

The study endpoints include the analysis of the graft site via study procedures at different time points, the comparison of cotton rolling to centrifugation method of autologous fat grafting, as well as the correlation of cell behavior of the laboratory assays with clinical outcomes.

DETAILED DESCRIPTION:
Clinical use of autologous fat grafting in humans was described as early as 1893, when Neuber published his report of transferring multiple small particles of fat to fill a soft tissue depression. Over the past three decades, autologous fat grafting has become a common procedure in clinical plastic surgery, and is also employed by clinicians in other specialties. The refinement of liposuction techniques in the 1980's made it possible to harvest the adipose grafts with low risk and without the need for a significant incision. The liposuction aspirate could simply be reinjected at a different site. Specialized equipment has been developed for fat grafting and is commercially available from a number of sources. The American Society of Plastic Surgeons 2007 procedural statistics show that over 65,000 fat grafting procedures were performed in the United States (www.plasticsurgery.org) during the previous year.

Fat grafting may represent a superior method of facial reconstruction after severe trauma, but the results can be impacted by resorption of fat volume over time. The specific aims of the study are:

1. Assess facial appearance and soft tissue volume before and after autologous fat grafting using CT scans and 3D photography.
2. Assess cellular properties of the cells within the fat graft
3. Comparison of cotton rolling to centrifugation method of autologous fat grafting
4. Measure of quality of life in patients before and after autologous fat grafting using validated psychosocial measures.

Ten (10) subjects 18 years of age and older will be enrolled to this trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older and able to provide informed consent
* Who are post injury and/or post surgery (e.g. tx of aneurism, intercranial bleed, and tumor resections that do not involve radiation and would be analogous to trauma population requiring craniotomy) resulting in craniofacial volume defect which could be treated with a graft volume of between 5 and 150 cc of lipoaspirate
* Be at least 3 months post-injury or post-surgery (from trauma procedures) so that acute edema is resolved
* Volume defects are covered by intact skin and do not communicate with oral cavity or sinuses
* The three dimensional geometry of the volume defects would allow for treatment with lipoaspirate injection that in a manner that at least two distinct treated areas could be discerned on gross examination
* Willing and able to comply with follow up examinations, including radiographic studies

Exclusion Criteria:

* Age less than 18 years
* Inability to provide informed consent
* Craniofacial defects intended for treatment have open wounds or communicate with oral cavity or sinus (note: presence of such a defect in the setting of another defect(s) that meets treatment criteria will not exclude the patient from participating)
* Active infection anywhere in the body
* Diagnosed with cancer within the last 12 months and /or presently receiving chemotherapy or radiation treatment
* Known coagulopathy
* Pregnancy
* Subjects with an Axis I DSM-IV diagnosis (e.g., Schizophrenia, Bipolar disorder) who are found to be clinically (i.e. medically) unstable at baseline. Individuals who manifest either: 1) evidence of currently active alcohol or psychoactive drug abuse or dependence on the SCID interview, or 2) a GAF score of 40 or lower due to any acute psychiatric symptomatology (e.g. suicidality, psychosis, severe depression or mania) will be reviewed by the Co-I for Psychosocial Assessment with the PI for determination of possible medical instability. Final determination of medically unstable status will be made by the PI on the basis of overall medical status and appropriateness for medical procedures; the patient may be considered ineligible for study participation per the Physician's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Rubin, MD, Principal Investigator — Professor of Plastic Surgery at the University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
It is the Principal Investigator's intention to make stored samples and subject information de-identified available to secondary investigators (investigators not listed on the front page of this consent document) after all research study testing has been completed. These stored samples and associated subject information will not include subject identifiers.

REFERENCES:
- [Derived] Bourne DA, Bliley J, James I, Donnenberg AD, Donnenberg VS, Branstetter BF 4th, Haas GL, Radomsky E, Meyer EM, Pfeifer ME, Brown SA, Marra KG, Coleman S, Rubin JP. Changing the Paradigm of Craniofacial Reconstruction: A Prospective Clinical Trial of Autologous Fat Transfer for Craniofacial Deformities. Ann Surg. 2021 May 1;273(5):1004-1011. doi: 10.1097/SLA.0000000000003318. PMID 30985369

RESULTS

PARTICIPANT FLOW:
Groups:
- Cotton Rolling Fat Grafting: For the purpose of this study the fat grafting procedure is a research procedure. It is very important to note that this research procedure is not an experimental procedure. Fat grafting is a minimally invasive clinical procedure that has been widely used by plastic surgeons within reconstructive surgery for many years. Fat grafting is known as a filler providing an accurate means to restoring facial soft tissue structure.
  The processing of the fat graft material is done using a cotton rolling technique via a Tefla non-adherent gauze pad in a rolling technique that separates the aqueous and oil layers from the injected component.
Period: Overall Study
Arm/Group | Cotton Rolling Fat Grafting
Started | 15
Completed | 10
Not Completed | 5
Not completed — Physician Decision | 2
Not completed — Screen fail | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cotton Rolling Fat Grafting
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Soft Tissue Volume After Autologous Fat Grafting Using CT Scans.
Time Frame: Assessed at 7-21 days, 3 months, 9 months
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Cotton Rolling Fat Grafting
Number analyzed (Participants) | 10
milliliters
  7-21 days | 11.4 (6.6)
  3 months | 7.4 (4.9)
  9 months | 6.5 (4.7)

2. Primary Outcome: Facial Volume Appearance of Each Subject Was Evaluated by the Clinician at Screen, 7-21 Days, 3, and 9 Months Post-operative.
Description: Facial volume appearance is based on the established Facial Volume Appearance Scale (FVAS). The scale is from 1-3 where 1 indicates no improvement and 3 indicates noticeable improvement of facial volume appearance.
Time Frame: screen, 7-21 days, 3, and 9 months post-operative
Measure: Mean (Standard Deviation); unit: units on FVAS scale
Arm/Group | Cotton Rolling Fat Grafting
Number analyzed (Participants) | 10
units on FVAS scale
  screen | 1.0 (0.0)
  7-21 days | 2.6 (0.5)
  3 months | 2.2 (0.4)
  9 months | 2.2 (0.4)

3. Secondary Outcome: Assessment of Cellular Properties of the Cells Within the Fat Graft
Description: Properties will be assessed via flow cytometry to measure the percentage of ASCs (adipose stem cells) within the SVF (stromal vascular fraction) from the fat graft.
Time Frame: Assessed at time of operative procedure
Measure: Mean (Standard Deviation); unit: percentage of ASCs within the SVF
Arm/Group | Cotton Rolling Fat Grafting
Number analyzed (Participants) | 10
percentage of ASCs within the SVF | 27.9 (17.7)

ADVERSE EVENTS:
Time Frame: 7-21 days, 3 months, 9 months post-operatively.
Arm/Group | Cotton Rolling Fat Grafting
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cotton Rolling Fat Grafting (N=10)
Bruising (Surgical and medical procedures) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT02267187/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT02267187/ICF_001.pdf